CLINICAL TRIAL: NCT02039752
Title: Asan Medical Center Registry for Multivessel
Brief Title: Asan Multivessel Registry
Acronym: ASAN MV
Status: Recruiting | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2013-15
Record Dates: First submitted 2014-01-14; First posted 2014-01-20 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: Multivessel
MeSH Terms: conditions — Coronary Artery Disease | interventions — Therapeutics; Medically Underserved Area; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Multivessel: from 1995
  Interventions: Other: Treatment

INTERVENTIONS:
Other: Treatment
  Other Names: Medically; Surgically; Percutaneously

SUMMARY:
The purpose of this study is to evaluate long-term prognoses of patients with multivessel coronary disease treated medically or surgically or percutaneously in real world practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multivessel disease from 1995 in Asan Medical Center
* Age 19 and more

Exclusion Criteria:

* For prospective cohort, not agreeing to participate with written informed consent form

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multivessel disease from 1995 in Asan Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
composite event | 1year
  death, myocardial infarction, stroke, revascularization

SECONDARY OUTCOMES:
Death | 1year
Myocardial Infarction | 1year
Stroke | 1year
Revascularization | 1year
Angina symptom | 1year
Bleeding | 1year
Re-hospitalization | 1year
Stent thrombosis | 1year
  by ARC(Academic Research Consortium) category

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park J, Kim SH, Kim M, Lee J, Choi Y, Kim H, Kim TO, Kang DY, Ahn JM, Yoo JS, Kim HJ, Kim JB, Choo SJ, Chung CH, Park SJ, Park DW; Asan-Multivessel Registry Investigators. Impact of Optimal Medical Therapy on Long-Term Outcomes After Myocardial Revascularization for Multivessel Coronary Disease. Am J Cardiol. 2023 Sep 15;203:81-91. doi: 10.1016/j.amjcard.2023.06.083. Epub 2023 Jul 21. PMID 37481816
- [Derived] Kim TO, Kang DY, Ahn JM, Kim SO, Lee PH, Lee J, Kim JH, Kim HJ, Kim JB, Choo SJ, Chung CH, Lee JW, Park SJ, Park DW; Asan Medical Center-Multivessel Revascularization Registry Investigators. Prognostic Impact of Mildly Impaired Renal Function in Patients Undergoing Multivessel Coronary Revascularization. J Am Coll Cardiol. 2022 Apr 5;79(13):1270-1284. doi: 10.1016/j.jacc.2022.01.035. PMID 35361350
- [Derived] Kim TO, Ahn JM, Kang DY, Park H, Kim SO, Lee PH, Lee J, Kim JH, Jeong YJ, Yang Y, Hyun J, Kim HJ, Kim JB, Choo SJ, Chung CH, Lee JW, Park SJ, Park DW; Asan-Multivessel Registry Investigators. Long-Term Outcomes After Percutaneous Coronary Intervention With Second-Generation Drug-Eluting Stents or Coronary Artery Bypass Grafting for Multivessel Coronary Disease. Am J Cardiol. 2021 Dec 1;160:21-30. doi: 10.1016/j.amjcard.2021.08.047. Epub 2021 Oct 3. PMID 34610874